CLINICAL TRIAL: NCT05895188
Title: The Effect Of Virtual Reality Glasses Applied During Pap Smear On Anxiety, Pain And Patient Satisfaction: A Randomized Controlled Trial
Brief Title: The Effect Of Virtual Reality Glasses Applied During Pap Smear On Anxiety, Pain And Patient Satisfaction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Hacer Gülen Savaş, PhD, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DU-SBF-RS-01
Record Dates: First submitted 2022-12-10; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-05

CONDITIONS: Anxiety; Pain; Patient Satisfaction
Keywords: Papanicolaou Test; Virtual Reality
MeSH Terms: conditions — Anxiety Disorders; Pain; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: In the study, there are two groups, the virtual reality group in which virtual reality glasses were applied and the control group, which did not apply any intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: There are two groups in the study and the informed consent texts of these groups are different. In this way, the participants will not know which group they belong to. The randomization table of the study was made by an independent researcher, so the researcher would not know which patient was in which group. At the end of the research, data analysis will be done by an independent statistician, and the statistician will not know which patient's data belongs to which group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Before starting the process, participants will be informed about the study and their verbal and written consent will be obtained. Participants in the virtual reality group will be shown and introduced to virtual reality glasses before the procedure. After the woman goes to the examination table and takes the appropriate position for the pap smear procedure, virtual reality glasses will be put on the woman by the researcher. The selected video will be played until the Pap smear process is completed. (https://www.youtube.com/watch?v=6ud18oSuCiY&t=30s). When the Pap smear is finished, the glasses will be removed and the woman will be helped to get up from the examination table. In this process, no form will be filled until the participant woman gets dressed and takes the ready position. Thus, the privacy of women will be protected and there will be no violation of ethical rights.
  Interventions: Device: Virtual Reality Glasses
- Control Group (No Intervention): Verbal and written consent will be obtained from the participants before starting the procedure. No intervention will be applied to the participants in the control group. The forms that need to be filled before the procedure will be filled. With the help and guidance of the researcher, the woman will prepare, move to the examination table and take a position. After the Pap smear process is over, the participant woman will get off the examination table with the help of the researcher and get dressed. After the woman is ready after the procedure, she will go to the waiting room and fill out the forms.

INTERVENTIONS:
Device: Virtual Reality Glasses — From the beginning to the end of the procedure, women will watch the selected nature video.
  Arms: Virtual Reality Group

SUMMARY:
This research is a randomized controlled experimental study designed to determine the effect of video, which is watched by virtual reality glasses during the procedure, on anxiety, pain and patient satisfaction to women who have had pap smear test.

DETAILED DESCRIPTION:
Cervical cancer is the most important preventable gynecological cancer that can be diagnosed with early screening among female gynecological cancers. Today, cervical cancer has become an important public health problem (General Directorate of Public According to the data of the Global Cancer Observatory (GLOBOCAN), a subsidiary of the World Health Organization, 604,127 women were diagnosed with cervical cancer in 2020. With these new cases, cervical cancer ranked 4th worldwide in incidence and mortality. In Turkey, the incidence of cervical cancer ranks 3rd among gynecological cancers. In the world and in Turkey. The primary prevention of this cancer type, which has a high mortality rate in addition to its incidence rate, is the Human Papilloma Virus (HPV) vaccine. Secondary prevention includes early diagnosis with screening tests. Screening tests for the diagnosis of cervical cancer are pap smear test and HPV DNA test.

Thanks to the Pap smear screening test, the diagnosis can be made even if cervical cancer does not show any symptoms. In addition, preinvasive and invasive lesions of cervical cancer can be detected. Thanks to these features of the Pap smear test, lesions can be detected in the early period, the treatment process can be started early, and mortality and morbidity rates can be reduced. The Pap smear test is an easy-to-apply, inexpensive, reliable and easy-to-access screening test. It has been reported that regular pap smear test screening reduces the mortality and morbidity rate of cervical cancer by 70% in developed countries. It is recommended by the Ministry of Health that women over the age of 30 should have a pap smear test once every 5 years. It is recommended that screening be discontinued in women who have 3 consecutive negative tests or who are over 65 years old. Despite the recommendations and practices of the Ministry of Health, 20% of women in Turkey were screened within the scope of the screening program. Studies conducted in the national and international literature reveal many reasons why women do not have a pap smear test.

The primary reason why women do not have a pap smear test is gynecological examination. Women may experience anxiety and worry due to the speculum used during the gynecological examination, the fact that the procedure area is a private area, and the possibility of being diagnosed with cancer as a result of the test. In a study, it was found that 20.7% of women experienced moderate anxiety and 10.9% had high level anxiety before the gynecological examination. In another study, the state anxiety score of women who applied for a pap smear test was found to be high. Women may develop negative attitudes towards screening tests due to the anxiety they experience. For this reason, early diagnosis may miss the opportunity. Özcan et al. recommend that nurses provide supportive care to women during gynecological examination and reduce their anxiety.

Distraction method and pain and anxiety management are among the independent roles of nurses. There are many nursing practices that can be done to reduce the anxiety and pain feelings of patients. Virtual reality application is also used as one of these applications. With the developing technology, virtual reality applications have started to be applied as a distraction technique. Created as a result of combining three-dimensional and interactive graphics prepared in virtual reality computer environments with various programs in the computer environment, it has been defined as technologies that draw users directly into a virtual world and create the feeling of being in the real world. The sensors placed in the virtual reality glasses detect the head movements of the user and act in sync with the virtual environment, allowing the individual to see the place where the individual turns his head in the virtual environment. Thanks to this feature of virtual reality glasses, people can make nature, underwater and museum tours. Virtual reality glasses create a feeling of being in a virtual environment. Thus, the person can completely move away from the environment. This feature of virtual reality applications is mostly used in the medical field. People are moving away from the medical environment they are in, they feel as if they are in the images being watched. In this way, their attention can be diverted and their anxiety levels can be reduced. As people focus on the images they see, pain signals reach the brain later and there is a decrease in pain sensation. Anxiety and pain can be reduced with virtual reality application during invasive procedures such as hysteroscopy, amniocentesis, curettage, embryo transfer. reduction studies have been carried out. In the study of Deo et al., qualitative interviews were conducted at the end of the virtual reality application. 85% of the participants stated that the virtual reality application removed them from the examination environment, thus they felt less pain and their anxiety decreased.

Studies using virtual reality during gynecological and obstetric diagnosis and treatment procedures have been found in the literature. In the available literature, no study has been found in which virtual reality is applied to women who will undergo pap smear test. With this study, it was aimed to increase patient satisfaction by reducing the pain and anxiety experienced during the pap smear screening test. In addition to this purpose, this study is important in terms of showing that virtual reality application, which is a product of developing technology, is adaptable and applicable to nursing care. It is thought that the health worker can also apply the procedure more easily, thanks to the reduction and relaxation of the anxiety of the woman during the procedure. As a result of the study, it is thought that if the pain and anxiety levels of women are reduced, the rates of having pap smear screening test will increase in the long run. In the study of Marashi et al., negative experiences during the first test were shown as one of the reasons why women did not have a pap smear test. It is thought that the negative experiences of women will be minimized by reducing the level of pain and anxiety. It is thought that the results of the research will contribute to the current literature.

ELIGIBILITY:
Inclusion Criteria:

* A sufficient level of education to understand study procedures and be able to communicate with site personnel
* Being in the age range of 30-65,
* To have Pap Smear test for the first time,
* Speaking Turkish and reading and writing,
* No vision and hearing problems,
* Not using glasses,
* Not a diagnosed psychiatric disease.

Exclusion Criteria:

* Having any physical or mental problems that may prevent communication
* To have a Pap Smear test before.
* Removing virtual reality glasses during the process
* Not filling the post -test form after the procedure.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Being a woman to have a pap smear test
Enrollment: 60 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-10-17 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Anxiety Level | 15 minutes
  Anxiety will be measured with the Visual Analog Scale (VAS-Anxiety). The Anxiety Visual Analog Scale includes numbers from 0 to 10, the higher the number marked, the higher the level of anxiety felt.Anxiety level will be measured twice, before and after the procedure.
State Anxiety Level | 15 minutes
  Anxiety level after the procedure will be measured with the State Anxiety Inventory (STAI I). The state anxiety scale measures the level of anxiety felt at the moment. It consists of 20 items, scores range from 20-80. The higher the score, the higher the level of anxiety felt. state anxiety level will be measured once after the pap smear process is completed.

SECONDARY OUTCOMES:
Pain Level | 15 minutes
  It will be measured with the Visual Analog Scale (VAS). The visual analog scale includes numbers 1-10, as the marked number increases, the level of pain felt increases.
patient satisfaction level | 15 minutes
  It will be measured by the evaluation form of numerical patient satisfaction. It is formed in a single -item likert type. It is scored between 1-5 points. As the score increases, the level of satisfaction for the Pap Smear test increases.
virtual reality application satisfaction level | 15 minutes
  Satisfaction with Virtual Reality will be measured with the Evaluation Form. It was created in a 5-point likert type. It consists of 12 items. The highest satisfaction score is 40 points because it also includes negative statements. As the score increases in the range of 40-75 points, satisfaction decreases.

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÜLEN SAVAŞ, PhD, Principal Investigator — Duzce University
Locations (1):
- Düzce General Directorate of Public Health Cancer Early Diagnosis Screening and Training Center, Düzce, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No